CLINICAL TRIAL: NCT00587821
Title: Peptide Profiles of Women Undergoing Breast Biopsy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 06-003
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: The first 250 samples will be used as a training set and results of these breast biopsies (benign or malignant) will be used to determine the peptide profile characteristic of a diagnosis of breast cancer on biopsy.
  Interventions: Other: Blood draw
- 2: The predictive capacity of this profile will then be prospectively assessed using the next 250 samples, which will serve as a validation set. Subjects who are candidates for enrollment on cohort B of this study (metastatic disease)
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Peptide profiles from blood samples of all subjects will be determined by mass spectrometric analysis.

SUMMARY:
This study is being done to learn about blood proteins. We want to see if the blood proteins in women whose biopsies show breast cancer are different from the blood proteins in women whose biopsies do not show breast cancer. The goal of this study is to develop a blood test than can help detect breast cancers when they are very small and easy to cure.

DETAILED DESCRIPTION:
Despite currently available screening techniques, only 63% of breast cancer cases are diagnosed at a localized stage, for which the 5-year survival rate exceeds 95% (1). Advances in breast imaging are occurring, but further efforts to detect breast cancer at an early stage would be beneficial. Recently, new technologies which use mass spectrometric analysis to characterize the overall pattern of peptide expression in the serum or plasma have been developed. Preliminary studies have suggested that peptide profiles can be used to differentiate cancer patients from those without cancer for a variety of malignancies including breast cancer. If mass spectrometric analysis is able to detect differences in peptide profiles between early stage breast cancers and normal controls, this technique could be developed as a screening modality.

The objective of the present study which is entitled "Peptide Profiles of Women Undergoing Breast Biopsy" is to determine whether the diagnosis of malignancy on breast biopsy is associated with a specific serum or plasma peptide profile which can be distinguished from the peptide profile associated with benign diagnoses on breast biopsy. To accomplish this, blood samples will be collected from 500 women undergoing breast biopsy and 100 women with metastatic disease. Samples will be obtained prior to the biopsies and analyzed by mass spectrometry. Residual material will be shared with investigators of the National Cancer Institute Clinical Proteomics Technology Assessment Consortium.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ or = to 18

Cohort A: Biopsy Cohort:

* Referred by a healthcare provider for breast biopsy
* No prior history of invasive breast cancer OR of ductal carcinoma in situ
* No prior history of other malignancies within 5 years except cervical dysplasia, squamous cell carcinoma of the skin or basal cell carcinoma of the skin Cohort B: Metastatic Disease Cohort - Diagnosis of stage IV breast cancer

Exclusion Criteria:

* Male
* Age < 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Other potential subjects will be informed of the study by her treating professional at the time she is told of the need for a biopsy. Lists of patients scheduled for biopsy will be reviewed by study personnel on a weekly basis.
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To identify the peptide profile associated with a diagnosis of malignancy on breast biopsy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org